CLINICAL TRIAL: NCT02127840
Title: Influence of Synacthen Infusion on the Results of Adrenal Venous Sampling in Patient With Primary Aldosteronism
Acronym: ISIRA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Miroslav Solar, Principal Investigator, Charles University, Czech Republic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PAAVS1143
Record Dates: First submitted 2014-04-25; First posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Primary Aldosteronism
Keywords: primary aldosteronism; adrenal adenoma; arterial hypertension
MeSH Terms: conditions — Hyperaldosteronism; ACTH Syndrome, Ectopic; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Synacthen (Experimental): Synacthen infusion during adrenal venous sampling
  Interventions: Drug: Synacthen infusion during adrenal venous sampling
- Without Synacthen (No Intervention): Adrenal venous sampling without Synacthen

INTERVENTIONS:
Drug: Synacthen infusion during adrenal venous sampling — Adrenal venous sampling during Synacthen infusion
  Arms: Synacthen

SUMMARY:
The project is aimed to determine the value of synacthen infusion on the results of adrenal venous sampling in patients examined for primary aldosteronism

DETAILED DESCRIPTION:
We aim to compare the results of adrenal venous sampling performed without and during synacthen infusion.

ELIGIBILITY:
Inclusion Criteria: Confirmed primary aldosteronism

Exclusion Criteria: Inability to undergo unilateral adrenalectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
To verify whether Synacthen infusion may influence the results of adrenal venous sampling in patients with primary aldosteronism | End of clinical examination procedure, i.e. within 4 week after adrenal venous sampling is performed.

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Ceral, MD, Study Chair — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia